CLINICAL TRIAL: NCT04247256
Title: An Open-label Phase II Prospective Clinical Trial to Investigate Safety, Tolerability, Maximum Tolerated Dose and Anti-tumor Effect for SCO-101 in Combination With FOLFIRI as a Safe and Efficient Treatment Modality in Metastatic or Advanced Colorectal Cancer (mCRC) Patients With Acquired FOLFIRI Resistant Cancer Disease.
Brief Title: A Phase 2 Trial of SCO-101 in Combination With FOLFIRI for Patients With Metastatic Colorectal Cancer (mCRC) With Acquired Resistance to FOLFIRI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scandion Oncology A/S (Industry)
Collaborators: TFS Trial Form Support (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCO101-001
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal; cancer; resistant; FOLFIRI; metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — IFL protocol

STUDY DESIGN:
Intervention Model Description: This is a multi-center, open label, dose escalation, Phase 2 study of SCO-101 in combination with FOLFIRI in up to 50 mCRC patients.
  Cohorts of FOLFIRI-resistant mCRC patients will be treated with SCO-101 in combination with FOLFIRI . Patients to be enrolled should previously have had either complete response (CR), partial response (PR), or stable disease (SD) (>16 weeks) on FOLFIRI.
  The study is separated in two parts. Part 1 is a dose escalation part with a standard 3+3 design, designed to evaluate the safety and toxicity of the combination of SCO-101 and FOLFIRI, and to identify the maximum tolerated dose (MTD). A maximum of 5 cohorts have been planned. Starting dose of SCO-101 is 150 mg (cohort 1) and maximum dose is 350 mg (cohort 5).
  Part 2 is the efficacy part, where patients are treated with the MTD dose identified in the first part and evaluated for efficacy and safety of the combination SCO-101 plus FOLFIRI.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): SCO-101 in combination with FOLFIRI
  Interventions: Drug: FOLFIRI Protocol; Drug: SCO-101

INTERVENTIONS:
Drug: FOLFIRI Protocol — FOLFIRI standard treatment on day 5 to 7 (both days included) of a 14 day period. repeated bi-weekly
Drug: SCO-101 — Investigational Medicinal Product, oral tablet administered on day 1 to 6 (both days included) of a 14 day period. repeated bi-weekly

SUMMARY:
This study evaluates the combination of SCO-101 to FOLFIRI for the treatment of metastatic colorectal cancer patients who have developed resistance to FOLFIRI treatment. The study is divided in two parts, where the first part evaluates the safety and toxicity of increasing doses of SCO-101 in combination with FOLFIRI at the same dose as the patient has previously developed resistance to. The second part of the study evaluates the safety and efficacy of the combination of FOLFIRI and SCO-101 at the dose level established in the first part.

DETAILED DESCRIPTION:
This is a multi-center, open label, dose escalation, Phase 2 study of SCO-101 in combination with FOLFIRI in up to 50 mCRC patients. All patients included have previously had effect from treatment with FOLFIRI, but have now progressed (i.e. treatment failure due to acquired resistance).

FOLFIRI is a key anti-cancer chemotherapeutic combination in the treatment of several solid tumor cancers, e.g. colorectal cancer. Cancer resistance to FOLFIRI exposure is a well known phenomenon and can often be attributed to upregulation of cellular efflux pumps, e.g. ATP-Binding Cassette (ABC)G2 and ABCB1, involved in the efflux of the chemotherapeutic agents from the cancer cells and resulting in treatment failure.

SCO-101 is an inhibitor of ATP-Binding Cassette (ABC) efflux pumps and SRPK1 kinase which is responsible for phosphorylation of splicing factors, a key element involved in tumour growth.

The combination of SCO-101 with FOLFIRI is expected to inhibit the active efflux of chemotherapy molecules from the cancer cell thereby re-sensitizing it to the chemotherapeutic agents.

ELIGIBILITY:
Inclusion Criteria: Subjects are required to meet all of the following criteria for enrollment into the applicable stage (stage 1, stage 2 or stage 3) of the study:

1. Ability to understand and willingness to provide written informed consent before any trial-related activities.
2. Age 18 years or older.
3. Histologically verified colorectal adenocarcinoma.
4. Non-resectable mCRC in patients A. Stage 1 only: with or without known BRAF, KRAS or repair enzyme mutations. B. Stage 2 and stage 3 only: without known BRAF, KRAS or repair enzyme mutations
5. A. Stage 1 only: Documented progressive disease on FOLFIRI treatment regimen (with or without antiangiogenetic and EGFR inhibitory biological treatment).

   B. Stage 2 and stage 3 only: Documented progressive disease with a prior benefit (SD for more than 16 weeks, or CR or PR) on FOLFIRI treatment regimen (with or without antiangiogenetic and EGFR inhibitory biological treatment).
6. Maximum reduction of 33% in prior dose of FOLFIRI.
7. No indication for treatment with an oxaliplatin-containing treatment regimen. The patient may have received oxaliplatin treatment after treatment with FOLFIRI.
8. A. Stage 1 only: Evaluable disease by CT scan or MRI. B. Stage 2 and stage 3 only: Measurable disease by CT scan or MRI, according to RECIST. 1.1.
9. Performance status of ECOG ≤ 1.
10. Recovered to Grade 1 or less from prior surgery or acute toxicities of prior radiotherapy or treatment with cytotoxic or biologic agents.
11. ≥ 2 weeks must have elapsed since any prior surgery.
12. Adequate conditions as evidenced by the following clinical laboratory values:

    * Absolute neutrophils count (ANC) ≥ 1.5 x 109/L
    * Haemoglobin ≥ 6.0 mmol/L
    * Platelets ≥ 100 x 109 /L
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN*
    * Total serum bilirubin ≤ 1.0 ULN**
    * Alkaline phosphatase ≤ 2.5 x ULN*
    * Creatinine ≤ 1.5 ULN
    * eGFR within normal limits.
    * Adequate blood clothing function as defined by the International Normalized Ratio (INR) ≤ 1.2;
13. Life expectancy equal to or longer than 3 months.
14. Sexually active males and females of child-producing potential must use highly effective contraception (intrauterine devices, hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release)) for the study duration and at least 6 months after the last dose of study drug.
15. Signed informed consent.

    * AST is not mandatory. In case of known liver metastases with ALT and AST ≤ 5 x ULN and/or alkaline phosphatase ≤ 5 x ULN: Patients who do not conform to the transaminase and/or alkaline phosphatase inclusion criteria, but who by the PI are considered in good PS and otherwise eligible for inclusion, and where the transaminase and/or alkaline phosphatase levels are considered elevated due to other reasons than deteriorated lever capacity, may be considered for inclusion based on conferred agreement between PI and sponsor.

      * Unconjugated bilirubin may be measured as the difference between total bilirubin and conjugated bilirubin.

Exclusion Criteria: Subjects meeting any of the following criteria will be excluded from enrollment:

1. Concurrent chemotherapy, radiotherapy, or other investigational drug except non-disease related conditions (e.g. insulin for diabetes) during study period.
2. Malabsorption syndrome or previous surgeries with resection of the stomach or small intestine, whereby absorption of SCO-101 may be affected. This includes patients with ileostomy.
3. Difficulty in swallowing tablets.
4. Clinical symptoms of CNS metastases requiring steroids.
5. Any active infection requiring parenteral or oral antibiotic treatment.
6. Known HIV positivity.
7. Known active hepatitis B or C.
8. Clinical significant (i.e. active) cardiovascular disease:

   * Stroke within ≤ 6 months prior to day 1
   * Transient ischemic attach (TIA) within ≤ 6 months prior to day 1
   * Myocardial infarction within ≤ 6 months prior to day 1
   * Unstable angina
   * New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF)
   * Serious cardiac arrhythmia requiring medication
9. Mental status is not fit for clinical study or CNS disease including symptomatic epilepsy.
10. Other medications or conditions that in the Investigator's opinion would contraindicate study participation of safety reasons or interfere with the interpretation of study results. Other severe medical conditions, including serious heart disease, unstable diabetes, uncontrolled hypercalcemia, clinically active infections or previous organ transplants. Participation in another clinical trial with experimental medication within 30 days prior to registration.
11. Known hypersensitivity to irinotecan, 5-FU or capecitabine
12. Pregnant women or women who are breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of combination of SCO-101 and FOLFIRI | 4 cycles (each cycle is 2 weeks)
  Safety and tolerability by assessing the number, frequency, and severity of adverse events (AEs) collected from the time of first treatment until four weeks after end of treatment to evaluate safety of SCO-101 in combination with FOLFIRI determined according to CTCAE version 5.0
Maximum Tolerated Dose | 1 cycle (each cycle is 2 weeks)
  Maximum tolerated dose (MTD) by evaluation of dose-limiting toxicities (DLTs) of SCO-101 in combination with FOLFIRI evaluated by CTCAE v. 5.0 (part 1 only)
Objective Response Rate | 4 cycles (each cycle is 2 weeks)
  Objective response rate (ORR) defined as CR and PR using the RECIST v. 1.1

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Start of treatment to first objective sign of progression, assessed up to 100 months
  Progression free survival (PFS) defined as time in months from the date of first study treatment to the date of disease progression or death from any cause, whichever comes first.
Duration of Response | From first response to progression, assessed up to 100 months
  Duration of response (from first response to progression)
Duration of Response compared to prior Duration of response | From first response to progression, assessed up to 100 months
  Duration of response (DOR) after administration of SCO-101 compared to DOR from patients initial FOLFIRI treatment regimen (without SCO-101).
Overall Survival | Up to 2 years
  Overall survival (OS) defined as time in months from the date of first study treatment to the date of death;
Clinical Benefit Rate | from benefit (CR, PR or SD > 16 weeks) to progression, assessed up to 100 months
  Clinical benefit rate (CBR) defined as the number of patients obtaining CR, PR, or SD > 16 weeks according to RECIST v.1.1.
Pharmacokinetic profile of SCO-101 in combination with FOLFIRI | First week of administration (study part 1 only)
  Pharmacokinetic profile of SCO-101 in blood samples
ctDNA | First 4 cycles of treatment (each cycle is 2 weeks) (study part 2 only)
  Change in ctDNA from baseline (prior first dose of SCO-101) until first CT scan
Biomarker UGT1A1 | Baseline (pre-treatment (all study parts))
  Evaluation of Selected UGT1A1 polymorphism in a pre-treatment blood sample
Biomarker IndiTreat(TM) | Baseline (pre-treatment tumor biopsy (study part 2 only))
  Efficacy of IndiTreat® to predict clinical response to SCO-101 treatment in combination with FOLFIRI from a tumor biopsy sample.
Biomarkers ABCG2, ABCB1, SRPK1 | Baseline (Pre-treatment biopsy (study part 2 only))
  Efficacy of molecular biomarkers ABCB1/ABCG2/SRPK1 determined by immunohistochemistry to predict clinical response to SCO-101 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Hagen Vasehus Schou, MD, Principal Investigator — Herlev and Gentofte Hospital
Locations (12):
- Denmark (6):
  - Aalborg Universitetshospital - Region Nordjylland, Aalborg
  - Herlev Hospital, Herlev
  - Hillerød Hospital, Hillerød
  - Sjællands Universitetshospital, Roskilde, Roskilde
  - Sygehus Sønderjylland, Sønderborg
  - Vejle Sygehus, Vejle
- Germany (3):
  - Charité, Berlin
  - Catholic Hospital Bochum - St. Josef-Hospital, Bochum
  - University Hospital Of Ulm, Ulm
- Spain (3):
  - Hospital de la Santa Creu in Sant Pau, Barcelona
  - Hospital Universitario Valle de Hebrón, Barcelona
  - Hospital Clínico Universitario in Valencia, Valencia